CLINICAL TRIAL: NCT02973815
Title: New Ulm at HOME (Healthy Offerings Via the Mealtime Environment), NU-HOME
Acronym: NU-HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Allina Health System (Other); Minneapolis Heart Institute Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1509S78583; 1R01HL123699 (NIH)
Record Dates: First submitted 2016-11-08; First posted 2016-11-25 (Estimated); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Obesity, Childhood; Physical Activity; Food Intake; Rural Health
Keywords: family meals; home food availability
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NU-HOME Intervention (Experimental): Participants randomized to the intervention condition will receive the NU-HOME family intervention program that includes group sessions with other families focused on nutrition education, cooking skills, and physical activity. The intervention program also includes individual goal setting phone calls with parents and online, complementary materials.
  Interventions: Behavioral: NU-HOME Intervention
- Delayed Intervention (No Intervention): Participants randomized to the delayed intervention condition will not receive any educational materials or training until after the final data collection. Once all data collection is completed, they will receive a shortened version of the NU-HOME intervention program that was offered to the intervention families.

INTERVENTIONS:
Behavioral: NU-HOME Intervention — The NU-HOME family intervention program consists of seven monthly group sessions, individual goal setting calls and online materials to support the sessions. The intervention focuses on promoting healthful family meals where parents and children cook and eat together, healthful home food and physical activity environments, and being active together as a family.
  Arms: NU-HOME Intervention

SUMMARY:
The goal of the proposed project is to see if an innovative family-based intervention can reduce childhood obesity by actively engaging the whole family in promoting healthy behaviors in the home. In addition, the project will also examine how the NU-HOME family intervention influences children's dietary intake, availability of healthy and unhealthy foods in the home and served at meals and snacks, physical activity as a family, and child screen time (TV, game systems). The study will build upon a similar project conducted in an urban area and translate the lessons learned and adapt the program for a rural community.

DETAILED DESCRIPTION:
Childhood obesity is a serious public health problem. Although previous environmental approaches to obesity prevention show some promise, most studies have not shown excess weight gain reductions. Moreover, few childhood obesity prevention studies significantly engage parents or focus on the home environment, which is essential to promote healthy behaviors at home. Children in rural communities are particularly vulnerable regarding increased risk for obesity; thus, successful programs that engage families in rural communities to prevent excess weight gain are critical. The proposed research project, New Ulm at Home (NU-HOME), is a unique collaboration between leaders in a rural community (New Ulm, Minnesota) and successful academic obesity researchers. The residents of New Ulm are poised for and are requesting interventions to promote healthful behavior change, particularly for youth. In conjunction with our many community stakeholder groups, the objective of the proposed research is to test the effectiveness of the NU-HOME program, a 7-month, family-based health promotion intervention to prevent excess weight gain (assessed via BMI z-score) among 7-10 year old children (n=114) in the New Ulm rural community. The intervention program is based on Social Cognitive Theory and a socio-ecological framework and will focus on novel health promotion components to prevent childhood obesity, including: 1) promoting regular meals in which family members cook and eat together (i.e., family meals), 2) promoting nutritionally-sound and appropriately-portioned snacks and meals, 3) reducing sedentary behavior, particularly screen time in the home setting, and 4) promoting physical activity through collaboration with community partners. The NU-HOME study is designed in four stages, including substantial formative work between the academic and community partners, a two-arm randomized controlled trial (RCT; intervention and wait-list control), and two activities to facilitate sustainability (delayed intervention delivery for control group participants and dissemination). A community-based participatory research (CBPR) approach will be used to adapt an existing program, HOME Plus that was piloted and shown to be effective in urban communities. The NU-HOME program has high translation potential and is likely to be immediately useful to rural families of school-age children because it will be tested in a real-world setting in collaboration with engaged, knowledgeable and influential community partners.

ELIGIBILITY:
Inclusion Criteria:

* child between the ages of 7-10 who lives with the target adult at least 50% of the time
* parent/guardian must be the primary-meal preparing parent/guardian

Exclusion Criteria:

* planning to move out of the area in the next 6 months
* medical condition that would prevent family from participating in group sessions

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayne A Fulkerson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, School of Nursing, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Helgeson E, Horning ML, Elgesma KM, Kubik MY, Fulkerson JA. Food Insecurity and Changes in Diet Quality and Body Mass Index z-Scores Among Elementary School Students. Child Obes. 2024 Oct;20(7):508-516. doi: 10.1089/chi.2023.0185. Epub 2024 Mar 28. PMID 38546529
- [Derived] Horning ML, Friend S, Freese RL, Barr-Anderson DJ, Linde JA, Sidebottom A, Sommerness SA, Fulkerson JA. Parent Weight, Diet, Active Living, and Food-Related Outcomes of the Family-Focused:NU-HOME Randomized Controlled Trial: NU-HOME Randomized Controlled Trial. J Acad Nutr Diet. 2023 May;123(5):751-760.e1. doi: 10.1016/j.jand.2022.10.009. Epub 2022 Oct 13. PMID 36244610
- [Derived] Linde JA, Horning Dehmer ML, Lee J, Friend S, Flattum C, Arcan C, Fulkerson JA. Associations of parent dietary role modeling with children's diet quality in a rural setting: Baseline data from the NU-HOME study. Appetite. 2022 Jul 1;174:106007. doi: 10.1016/j.appet.2022.106007. Epub 2022 Mar 21. PMID 35331787
- [Derived] Fulkerson JA, Horning M, Barr-Anderson DJ, Sidebottom A, Linde JA, Lindberg R, Friend S, Beaudette J, Flattum C, Freese RL. Weight outcomes of NU-HOME: a randomized controlled trial to prevent obesity among rural children. Int J Behav Nutr Phys Act. 2022 Mar 19;19(1):29. doi: 10.1186/s12966-022-01260-w. PMID 35305674
- [Derived] Horning ML, Friend S, Lee J, Flattum C, Fulkerson JA. Family Characteristics Associated with Preparing and Eating More Family Evening Meals at Home. J Acad Nutr Diet. 2022 Jan;122(1):121-128. doi: 10.1016/j.jand.2021.07.002. Epub 2021 Aug 13. PMID 34399976
- [Derived] Fulkerson JA, Horning ML, Barr-Anderson DJ, Linde JA, Sidebottom AC, Lindberg R, Friend S, Flattum C, Freese RL. Universal childhood obesity prevention in a rural community: Study design, methods and baseline participant characteristics of the NU-HOME randomized controlled trial. Contemp Clin Trials. 2021 Jan;100:106160. doi: 10.1016/j.cct.2020.106160. Epub 2020 Sep 28. PMID 33002598
- [Derived] Martin CL, Kramer-Kostecka EN, Linde JA, Friend S, Zuroski VR, Fulkerson JA. Leveraging Interdisciplinary Teams to Develop and Implement Secure Websites for Behavioral Research: Applied Tutorial. J Med Internet Res. 2020 Sep 23;22(9):e19217. doi: 10.2196/19217. PMID 32965234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 228 participants representing 114 parent/child dyads were recruited in 2 cohorts (summers of 2017 and 2018)
Period: Post Intervention
Arm/Group | NU-HOME Intervention | Delayed Intervention
Started | 116 (58 parent/child dyads) | 112 (56 parent/child dyads)
Completed | 108 (54 parent/child dyads) | 88 (44 parent/child dyads)
Not Completed | 8 | 24
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 7 | 24
Period: Follow-up
Arm/Group | NU-HOME Intervention | Delayed Intervention
Started | 108 (54 parent/child dyads) | 88 (44 parent/child dyads)
Completed | 106 (53 parent/child dyads) | 88 (44 parent/child dyads)
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: 114 parent/child dyads
Groups:
- Total: Total of all reporting groups
Arm/Group | NU-HOME Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 116 | 112 | 228
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Mean age is reported separately for the child participant and the parent participant.
  years
    Child mean age: number analyzed (Participants) | 58 | 56 | 114
    Child mean age | 9.0 (1.0) | 9.0 (1.1) | 9.0 (1.0)
    Parent mean age: number analyzed (Participants) | 58 | 56 | 114
    Parent mean age | 37.8 (5.0) | 37.8 (5.6) | 37.8 (5.3)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Child and parent data are reported separately
  Participants
    Child sex: number analyzed (Participants) | 58 | 56 | 114
    Child sex: Female | 32 | 35 | 67
    Child sex: Male | 26 | 21 | 47
    Parent sex: number analyzed (Participants) | 58 | 56 | 114
    Parent sex: Female | 57 | 54 | 111
    Parent sex: Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Parent and child data reported separately
  Participants
    Child Hispanic: number analyzed (Participants) | 58 | 56 | 114
    Child Hispanic | 4 | 4 | 8
    Parent Hispanic: number analyzed (Participants) | 58 | 56 | 114
    Parent Hispanic | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Parent and child data reported separately
  Participants
    Child: number analyzed (Participants) | 58 | 56 | 114
    Child: Black, Indigenous, Person of Color | 6 | 2 | 8
    Child: White | 52 | 54 | 106
    Parent: number analyzed (Participants) | 58 | 56 | 114
    Parent: Black, Indigenous, Person of Color | 2 | 2 | 4
    Parent: White | 56 | 54 | 110
Region of Enrollment [Number; unit: participants]
  United States | 116 | 112 | 228

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Body Mass Index (BMI) Z-score
Description: Trained study staff will measure weight and height to calculate body mass index (BMI) then adjust for the child's age and sex to get BMI percentiles and z-scores. A Z-score of 0 represents the population mean with a z-score above zero indicating BMI above the population mean and a negative z-score indicating values below the population mean.
Time Frame: Post intervention (9 months after baseline)
Population: 102 post intervention BMI z-scores
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 56 | 46
z-score | 0.69 (1.00) | 1.03 (0.89)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; This was adjusted for the baseline BMI-Z score, child sex, baseline child age, and economic assistance; Test type: Other; p = 0.342, Regression, Linear; Mean Difference (Final Values) = -0.062, 95% CI 2-sided [-0.194 to 0.067], Standard Error of Mean 0.065

2. Secondary Outcome: Change in Home Availability of Fruits
Description: Participants will report the number of fruits available in their home using the Home Food Inventory.
Time Frame: Post intervention (9 months after baseline)
Population: 94 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: fruits
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 52 | 42
fruits | 1.87 (3.62) | 0.57 (4.27)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline HFI Fruit value, and economic assistance status; Test type: Other; p = 0.09, Regression, Linear; Mean Difference (Net) = 1.25, 95% CI 2-sided [-0.20 to 2.71], Standard Error of Mean 0.73104

3. Secondary Outcome: Change in Home Availability of Vegetables
Description: Participants will report the number of vegetables available in their home using the Home Food Inventory.
Time Frame: Post Intervention (9 months after baseline)
Population: 94 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: vegetables
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 52 | 42
vegetables | 0.52 (3.37) | -0.76 (2.77)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline HFI Vegetable value, and economic assistance status; Test type: Other; p = 0.047, Regression, Linear; Mean Difference (Net) = 1.23, 95% CI 2-sided [0.02 to 2.44], Standard Error of Mean 0.61

4. Secondary Outcome: Change in the Quality of Food and Beverages Served at Family Meals
Description: Participants will report details of food offerings at 7 days of evening meals using the Evening Meal Screener and the quality will be assessed by using a healthfulness score that combines multiple aspects of the meal into a single score. We created the Healthfulness of the Evening Meal Scale which has a range of (-4 to 11) where higher values represent a better outcome.
Time Frame: Post intervention (9 months after baseline)
Population: 92 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 49 | 43
units on a scale | 0.18 (0.96) | -0.19 (1.22)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline healthfulness score and economic assistance status; Test type: Other; p = 0.019, Regression, Linear; Mean Difference (Net) = 0.48, 95% CI 2-sided [0.08 to 0.88], Standard Error of Mean 0.20

5. Secondary Outcome: Change in Dietary Intake of Vegetables
Description: Child dietary intake will be assessed using mean number of servings of vegetables from two 24-hour dietary recalls
Time Frame: Post intervention (9 months after baseline)
Population: 98 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: vegetables
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 54 | 44
vegetables | -0.27 (0.94) | -0.01 (0.69)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline vegetable intake, child age (baseline), parent education status (bachelors or higher vs lower); Test type: Other; p = 0.218, Regression, Linear; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.4 to 0.09], Standard Error of Mean 0.12

6. Secondary Outcome: Change in Child Dietary Intake of Fruit
Description: Child dietary intake will be assessed using mean number of servings of fruit from two 24-hour dietary recalls
Time Frame: Post intervention (9 months after baseline)
Population: 98 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: fruits
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 54 | 44
fruits | 0.28 (1.41) | -0.02 (0.95)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline fruit intake, child age (baseline), parent education status (bachelors or higher vs lower); Test type: Other; p = 0.066, Regression, Linear; Mean Difference (Net) = 0.37, 95% CI 2-sided [-0.03 to 0.77], Standard Error of Mean 0.2

7. Secondary Outcome: Change in Minutes of Child Moderate to Vigorous Physical Activity
Description: Children will wear an accelerometer (ActiGraph wGT3X-BT and GT3XP-BTLE models) for 7 days to measure their activity levels (e.g., minutes of Moderate-to-vigorous physical activity). Trained research staff distributed the monitors to child participants who wore the monitors on their right hip for 7 consecutive days during most waking hours, except when sleeping or doing water-related activities. Data were collected in 10-second epochs. Accelerometer data were analyzed with ActiLife software (version 6.9.1). Non-wear time was defined as any period of >60 minutes of consecutive zeros. To be included in the analyses, participants had to have a minimum of >8 hours of wear time on >3 days. Evenson cutpoints for children were used to classify physical activity intensites: sedentary (0-100), light (101-2295), moderate (2296-4011), and vigorous (>4012). Minutes engaged in Moderate to Vigorous Physical activity was analyzed.
Time Frame: Post intervention (9 months after baseline)
Population: 91 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: Minutes of physical activity
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 51 | 40
Minutes of physical activity | -1.06 (21.47) | -1.21 (23.01)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline MVPA, child age (baseline), and child sex; Test type: Other; p = 0.28, Regression, Linear; Mean Difference (Net) = -4.79, 95% CI 2-sided [-13.56 to 3.98], Standard Error of Mean 4.41

8. Secondary Outcome: Change in Child Screen Time Use
Description: Parents will report on child's daily minutes of screen time.
Time Frame: Post intervention (9 months after baseline)
Population: 98 change scores analyzed total (takes into account missingness in the predictors variables)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NU-HOME Intervention | Delayed Intervention
Number analyzed (Participants) | 54 | 44
minutes | -0.19 (0.89) | -0.20 (0.93)
Statistical Analysis 1: Comparison: NU-HOME Intervention vs Delayed Intervention; Adjusted for: baseline screentime, child age (baseline), and child sex; Test type: Other; p = 0.928, Regression, Linear; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.31 to 0.34], Standard Error of Mean 0.17

ADVERSE EVENTS:
Time Frame: from baseline to post intervention (9 months)
Arm/Group | NU-HOME Intervention | Delayed Intervention
All-Cause Mortality (participants affected / at risk) | 1/116 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/112
Other Adverse Events (participants affected / at risk) | 0/116 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT02973815/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT02973815/ICF_001.pdf